CLINICAL TRIAL: NCT00926601
Title: Prevalence and Clinical Significance of Co-infection of Mycoplasma Pneumoniae in Patients With Pulmonary Tuberculosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae-Joon Yim / Associate Professor, Seoul National University Hospital
Other Study IDs: H-0906-006-281
Record Dates: First submitted 2009-06-20; First posted 2009-06-23 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Mycoplasma Pneumonia; Pulmonary Tuberculosis
MeSH Terms: conditions — Pneumonia, Mycoplasma; Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sera of TB patient
Oversight: Data Monitoring Committee: No

SUMMARY:
Several case report showed that the co-infection of Mycoplasma pneumoniae in patients with pulmonary tuberculosis. The aim of this study is to elucidate the prevalence and its clinical significance of co-infection of Mycoplasma pneumonia in patients with newly diagnosed pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Bacteriologically or clinically diagnosed pulmonary TB
* Older than 17years

Exclusion Criteria:

* HIV positive
* Immune-compromized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonary tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-06

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea